CLINICAL TRIAL: NCT02959606
Title: SAFE (Sarpogrelate Anplone in Femoro-popliteal Artery Intervention Efficacy) Study : a Randomized Controlled Trial
Brief Title: SAFE (Sarpogrelate Anplone in Femoro-popliteal Artery Intervention Efficacy) Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung-Kee Min, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAFE
Record Dates: First submitted 2016-11-08; First posted 2016-11-09 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — sarpogrelate; Clopidogrel

ARMS (2):
- Sarpogrelate SR 300mg + ASA (Experimental): Sarpogrelate HCl SR 300mg is administrated to patients with PAD for 6 weeks after EVT for femoro-popliteal regions.
  Other Name: Anplone SR
  Interventions: Drug: Sarpogrelate SR 300mg
- Clopidogrel + ASA (Active Comparator): Clopidogrel is administrated to patients with PAD for 6 weeks after EVT for femoro-popliteal regions.
  Other Name: Plavix
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Sarpogrelate SR 300mg
  Other Names: Anplone SR
  Arms: Sarpogrelate SR 300mg + ASA
Drug: Clopidogrel
  Arms: Clopidogrel + ASA

SUMMARY:
After endovascular treatment (EVT) for peripheral artery disease (PAD), dual antiplatelet therapy (DAAT) of aspirin (ASA) and clopidogrel are currently drug of choice to prevent occlusion. Anplone SR®, controlled-released Sarpogrelate hydrochloride, has been introduced as an anti-platelet agent for the drug of PAD. The aim of this study was to compare the efficacy and safety of Anplone + aspirin and clopidogrel + aspirin in patients who underwent EVT for femoro-popliteal occlusive disease.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, >18 years old
2. Angiographically-confirmed significant femoro-popliteal (FP) stenosis or occlusion by atherosclerosis
3. Successful FP intervention; residual stenosis <30%
4. Without significant residual inflow disease; Intact iliac artery inflow (with or without intervention of iliac or below knee arteries)
5. patent outflow status; at least 1 arterial runoff in below knee arteries
6. All kind of fem-pop intervention including POBA, stent, DCB, DES for TASC A~ D

Exclusion Criteria:

1. At risk of hemorrhage, bleeding tendency or thrombophilia
2. Acute limb ischemia / inflammatory arterial disease
3. Contraindication or allergic to ASA, clopidogrel, Anplone
4. Medication of warfarin
5. Pregnancy, hepatic dysfunction, thrombocytopenia
6. Previous FP bypass or intervention
7. Impossible to stop clopidogrel before EVT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Restenosis rate (50%>) in 6 months by CT angiography | 6 months

SECONDARY OUTCOMES:
Target lesion restenosis(TLR) in 6 months | 6 months
Major bleeding complication | 6 months
Ipsilateral major amputation | 6 months
All-cause mortality | 6 months
All adverse events | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Seung-Kee Min,, Seoul, South Korea

REFERENCES:
- [Derived] Han A, Lee T, Lee J, Song SW, Lee SS, Jung IM, Kang JM, Gwon JG, Yun WS, Cho YP, Ko H, Park YJ, Min SK. A multicenter, randomized, open-labelled, non-inferiority trial of sustained-release sarpogrelate versus clopidogrel after femoropopliteal artery intervention. Sci Rep. 2023 Feb 13;13(1):2502. doi: 10.1038/s41598-023-29006-z. PMID 36781928
- [Derived] Ahn S, Lee J, Min SK, Ha J, Min SI, Kim SY, Cho MJ, Cho S; SAFE study investigators. SAFE (Sarpogrelate Anplone in Femoro-popliteal artery intervention Efficacy) study: study protocol for a randomized controlled trial. Trials. 2017 Sep 22;18(1):439. doi: 10.1186/s13063-017-2155-5. PMID 28938905